CLINICAL TRIAL: NCT01560195
Title: A Double-Blind, Placebo-Controlled, Multicenter, Randomized Study Evaluating the Prophylactic Use of Pegylated Recombinant Human Granulocyte Colony Stimulating Factor (rhG-CSF) on the Incidence of Neutropenia in Subjects With Advanced Non-Small-Cell Lung Cancer (NSCLC) Treated With Myelosuppressive Chemotherapy
Brief Title: A Study of Pegylated rhG-CSF as Support to Advanced Non-Small-Cell Lung Cancer (NSCLC) Patients Receiving Chemotherapy Receiving Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HHPG-19K -III-02
Record Dates: First submitted 2012-03-08; First posted 2012-03-22 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: NSCLC; Neutropenia; Febrile Neutropenia
Keywords: neutropenia; febrile neutropenia; chemotherapy
MeSH Terms: conditions — Neutropenia; Febrile Neutropenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pegylated rhG-CSF: 100µg/kg (Experimental): Staged III or IV NSCLC patients receiving chemotherapy and Pegylated rhG-CSF 100µg/kg
  Interventions: Drug: Pegylated rhG-CSF: 100µg/kg
- Pegylated rhG-CSF: 6mg (Experimental): Staged III or IV NSCLC patients receiving chemotherapy and pegylated rhG-CSF 6mg
  Interventions: Drug: Pegylated rhG-CSF: 6mg
- Placebo (Placebo Comparator): Staged III or IV NSCLC patients receiving chemotherapy and placebo in cycle 1 and rhG-CSF in cycle 2 to 4
  Interventions: Drug: placebo and rhG-CSF 5ug/kg/d

INTERVENTIONS:
Drug: Pegylated rhG-CSF: 100µg/kg — Patients were administered pegylated rhG-CSF 100 ug/kg once at the 3rd day of every chemotherapy cycle. Chemotherapy regimen: docetaxel 75 mg/m2; carboplatin area under curve[AUC] 5 or cisplatin 75 mg/m2.
  Arms: Pegylated rhG-CSF: 100µg/kg
Drug: Pegylated rhG-CSF: 6mg — Patients were administered pegylated rhG-CSF 6mg once at the 3rd day of every chemotherapy cycle. Chemotherapy regimen: docetaxel 75 mg/m2; carboplatin area under curve[AUC] 5 or cisplatin 75 mg/m2.
  Arms: Pegylated rhG-CSF: 6mg
Drug: placebo and rhG-CSF 5ug/kg/d — Patients receiving chemotherapy and placebo in cycle 1 and rhG-CSF 5ug/kg/d in cycle 2 to 4. Chemotherapy regimen: docetaxel 75 mg/m2; carboplatin area under curve[AUC] 5 or cisplatin 75 mg/m2.
  Arms: Placebo

SUMMARY:
Neutropenia is one of the most frequent adverse effects of chemotherapy, and the main factor to limit the dosage and the continuation of chemotherapy. A newly pegylated rhG-CSF was independently developed by JIANGSU HENGRUI Medicine Co., Ltd, China. Phase 1a, 1b and phase 2 trials have shown that pegylated rhG-CSF has decreased renal clearance, increased plasma half-life, and prolonged efficacy in compare with ﬁlgrastim. The purpose of this study is to determine the safety and effectiveness of pegylated rhG-CSF in preventing neutropenia following chemotherapy in patients with advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Investigator diagnosis of staged III or IV NSCLC
* Age 18 to 70 years
* ECOG performance status ≤ 1
* Chemotherapy naïve
* Body weight ≥ 45kg
* Hemoglobin ≥ 100g/L; white blood cell ≥ 4.0×109/L; absolute neutrophil count ≥1.5 × 109/L; platelet count ≥ 100 × 109/L
* Alanine transarninase ≤1.5×ULN; aspartate aminotransferase ≤1.5×ULN; serum creatinine ≤1.5×ULN; total bilirubin ≤1.5×ULN

Exclusion Criteria:

* History of systematic chemotherapy or radical radiation therapy
* Prior bone marrow or stem cell transplantation
* Received systemic antibiotics treatment within 72 h of chemotherapy
* Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Rate of grade 3/4 neutropenia in cycle 1 | 21 days
  the rate of ANC lower than 1.0 × 109/L

SECONDARY OUTCOMES:
Incidence of febrile neutropenia in cycle 1 | 21 days
  rate of ANC<1.0×109/L and auxiliary temperature>38.5℃
Rate of grade 3/4 neutropenia and incidence of febrile neutropenia in cycle 2 to 4 | Through 2 to 4 cycles
  The rate of ANC lower than 1.0 × 109 /L and rate of ANC<1.0×109/L and auxiliary temperature>38.5℃
Time to neutrophil recovery in the 4 chemotherapy cycles | Through 4 cycles
  After chemotherapy administration the time from the expected nadir until the patient's ANC increased to 2.0 × 109/L
Duration of 3/4 neutropenia in the 4 chemotherapy cycles | Through 4 cycles
  duration of ANC lower than 1.0 × 109/L
Objective response rate | Through 4 cycles
Progress free survival | Through 4 cycles
Overall survival | Through 4 cycles
Exploratory biomarkers research | Through 4 cycles
  Relationship between SNP and microRNA with myelosuppression and tumor response rate

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China